CLINICAL TRIAL: NCT02716857
Title: A Randomized Withdrawal, Double-blind, Placebo-controlled Phase 3 Trial to Evaluate the Efficacy and Safety of Egalet® Abuse-deterrent, Extended-release (ADER) Oxycodone Tablet, Egalet-002, in Patients With Moderate-to-Severe Chronic Low Back Pain
Brief Title: Efficacy and Safety of Egalet-002 in Patients With Moderate-to-Severe Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC-EG-302
Record Dates: First submitted 2016-03-08; First posted 2016-03-23 (Estimated); Last update posted 2018-03-05 (Actual); Status verified 2018-03

CONDITIONS: Moderate-to-severe Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxycodone extended-release (Experimental): Egalet ADER oxycodone tablet
  Interventions: Drug: Oxycodone extended-release
- Placebo of Oxycodone extended-release (Placebo Comparator): Egalet ADER oxycodone placebo tablet
  Interventions: Drug: Placebo of oxycodone extended-release

INTERVENTIONS:
Drug: Oxycodone extended-release
  Other Names: Egalet-002, Egalet ADER oxycodone
  Arms: Oxycodone extended-release
Drug: Placebo of oxycodone extended-release
  Arms: Placebo of Oxycodone extended-release

SUMMARY:
The purpose of this study is to determine the analgesic efficacy of Egalet-002 twice daily (BID) in patients with moderate-to-severe chronic low back pain

ELIGIBILITY:
Inclusion Criteria:

* Is an English-speaking man or woman between 18 and 75 years of age who has given written informed consent.
* Has a clinical diagnosis of moderate-to-severe low back pain (Quebec Task Force Class 1 to 3) for ≥6 months.
* Is opioid naïve (ie, taking <20 mg oxycodone/day or opioid equivalent) or is opioid experienced (ie, taking a dose between 20 and 240 mg [inclusive] oxycodone/day or opioid equivalent) for management of moderate-to-severe CLBP at least 14 days prior to screening and will, in the opinion of the investigator, continue to require opioid therapy (between 20 and 240 mg oxycodone/day, inclusive) for management of moderate-to-severe CLBP for the duration of the study.
* Has stable health, as determined by the investigator,
* If female, the patient is currently not pregnant, not breast-feeding, nor attempting to become pregnant (for 30 days before screening and throughout the duration of the study), or is of non-childbearing potential

Exclusion Criteria:

* Has cancer-related pain.
* Has a history of receiving >240 mg oxycodone (or equivalent) daily within 30 days before screening.
* Has a lumbar spinal infusion pump in use or used within 6 months before screening.
* Has clinically unstable cardiac disease (including atrial fibrillation, symptomatic bradycardia, unstable congestive heart failure, or active myocardial ischemia)
* Has positive urine drug toxicity screen for illegal or non-prescribed drugs
* Has current (or history of within the last 5 years prior to screening) drug dependence or substance abuse disorder according to Diagnostic and Statistical Manual of Mental Disorders, 5th Edition, Text Revision criteria (excluding nicotine).
* Has positive result for cannabinoids (even if legally prescribed).
* Has a history of attempted suicide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Measure of Average Pain Intensity past 24 hours, as measured by a 0-10 NPRS using eDiary collection daily at bedtime. | 16 weeks

SECONDARY OUTCOMES:
Efficacy: daily (past 24 hours) worst pain intensity score (WPI) | 16 Weeks
Safety: Incidence of TEAEs, including those leading to treatment withdrawal, and/or abnormal physical examination findings, vital signs measurements, ECGs, and clinical laboratory test results, related to treatment | 16 weeks

CONTACTS AND LOCATIONS:
Locations (74):
- United States (74):
  - Site 207, Birmingham, Alabama
  - Site 202, Mobile, Alabama
  - Site 253, Phoenix, Arizona
  - Site 260, Phoenix, Arizona
  - Site 268, Phoenix, Arizona
  - Site 282, Tucson, Arizona
  - Site 217, Anaheim, California
  - Site 280, Anaheim, California
  - Site 220, La Mesa, California
  - Site 235, Laguna Hills, California
  - Site 215, Long Beach, California
  - Site 238, Los Gatos, California
  - Site 262, Napa, California
  - Site 201, Oakland, California
  - Site 225, Sacramento, California
  - Site 231, San Diego, California
  - Site 237, San Diego, California
  - Site 221, Wildomar, California
  - Site 248, Boulder, Colorado
  - Site 228, Bradenton, Florida
  - Site 214, Clearwater, Florida
  - Site 270, Gainesville, Florida
  - Site 269, Inverness, Florida
  - Site 227, Jupiter, Florida
  - SIte 204, Lake Worth, Florida
  - Site 211, Miami Beach, Florida
  - Site 229, Miami Beach, Florida
  - Site 278, Plantation, Florida
  - Site 232, Port Orange, Florida
  - Site 264, Sarasota, Florida
  - Site 271, Winter Park, Florida
  - Site 223, Atlanta, Georgia
  - Site 212, Marietta, Georgia
  - Site 245, Boise, Idaho
  - Site 255, Chicago, Illinois
  - Site 222, Evansville, Indiana
  - SIte 236, West Des Moines, Iowa
  - Site 277, Overland Park, Kansas
  - Site 206, New Orleans, Louisiana
  - Site 224, Shreveport, Louisiana
  - Site 249, Pikesville, Maryland
  - Site 226, Boston, Massachusetts
  - Site 254, New Bedford, Massachusetts
  - Site 210, Bay City, Michigan
  - Site 244, Jackson, Mississippi
  - Site 234, Hazelwood, Missouri
  - Site 265, Omaha, Nebraska
  - Site 266, Princeton, New Jersey
  - Site 267, Somerset, New Jersey
  - Site 252, Albuquerque, New Mexico
  - Site 261, Kew Gardens, New York
  - Site 243, New York, New York
  - Site 233, Rochester, New York
  - Site 208, Williamsville, New York
  - Site 203, Charlotte, North Carolina
  - Site 213, Winston-Salem, North Carolina
  - Site 242, Winston-Salem, North Carolina
  - Site 276, Columbus, Ohio
  - Site 209, Franklin, Ohio
  - Site 259, Kettering, Ohio
  - Site 240, Toledo, Ohio
  - Site 239, Oklahoma City, Oklahoma
  - Site 279, Duncansville, Pennsylvania
  - Site 256, Jenkintown, Pennsylvania
  - Site 258, Lansdale, Pennsylvania
  - Site 205, Charleston, South Carolina
  - Site 247, Greenville, South Carolina
  - Site 251, Spartanburg, South Carolina
  - Site 218, Austin, Texas
  - Site 263, Hurst, Texas
  - Site 219, Richardson, Texas
  - Site 275, San Antonio, Texas
  - Site 241, Everett, Washington
  - Site 257, Spokane, Washington